CLINICAL TRIAL: NCT01774214
Title: Rapid Pediatric Fluid Resuscitation: a Randomized Controlled Trial Comparing the Efficiency of Two Provider-Endorsed Manual Fluid Resuscitation Techniques
Brief Title: Pediatric Fast Fluid Trial 2
Acronym: PFFT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Collaborators: Regional Medical Associates of Hamilton (Unknown)
Responsible Party: Principal Investigator, Melissa J Parker, MD, MSc, Assistant Professor of Pediatrics, McMaster Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-358
Record Dates: First submitted 2013-01-19; First posted 2013-01-23 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Resuscitation; Shock; Fluid Therapy; Pediatrics
Keywords: Resuscitation; Shock; Fluid Therapy; Pediatrics
MeSH Terms: conditions — Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): As this is a crossover trial, the study arms denote the order in which the two interventions are performed by the subject. In Arm A, subjects will perform the "Push-Pull Technique" of manual fluid resuscitation first, followed by the "Disconnect-Reconnect Technique" second. A washout period of at least 30 minutes between each of the two interventions will be observed.
  Interventions: Procedure: Push-Pull technique; Procedure: Disconnect-Reconnect Technique
- B (Experimental): As this is a crossover trial, the study arms denote the order in which the two interventions are performed by the subject. In Arm B, subjects will perform the "Disconnect-Reconnect Technique" of manual fluid resuscitation first, followed by the "Push-Pull Technique" second. A washout period of at least 30 minutes between each of the two interventions will be observed.
  Interventions: Procedure: Push-Pull technique; Procedure: Disconnect-Reconnect Technique

INTERVENTIONS:
Procedure: Push-Pull technique — Participants will administer 900 mL (60 mL/kg) of NS to a model of a 15 kg toddler in shock. The intervention is the mode of administration of the fluid. For the "Push-Pull Technique", the 7 cm catheter extension tubing will be connected to one of the three ports of a triple stopcock. A second of the 3 ports of the triple stopcock will be connected to an IV tubing set connected to a 1 L bag of NS. A 60 mL syringe will be connected to the third port of the triple stopcock. On verbal prompt, participants will "pull" fluid from the bag of NS by withdrawing the plunger of the 60 mL syringe, filling it with saline. They will then toggle the switch of the triple stopcock, so that it is "off" to the bag of NS and "open" to IV catheter extension tubing leading to the model. They will then depress the syringe plunger, administering the fluid to the model. These steps will be repeated until each participant believes that they have administered the requested volume of fluid to the model.
Procedure: Disconnect-Reconnect Technique — Participants will administer 900 mL (60 mL/kg) of NS to a model of a 15 kg toddler in shock. The intervention is the mode of administration of the fluid. For the "Disconnect-Reconnect Technique", the proximal end of the 7 cm catheter extension tubing will be capped with a needleless adapter. The subject will be provided with 60 mL syringes filled with NS, rapidly prepared in real time by an assistant. Syringes will be prepared by withdrawing NS from a 1 L bag via a Gambro Accessory spike. The subject will administer the requested volume of NS to the model by 1. grabbing one of the fluid-filled syringes 2. connecting the fluid-filled syringe to the needleless adapter, and 3. depressing the syringe plunger resulting in administration of the NS to the model. These steps will be repeated until the subject believes they have administered the requested volume of NS to the model. Testing will begin on verbal prompt. The subject and assistant will not be permitted to switch roles.

SUMMARY:
The purpose of this study is to determine which of two commonly used methods of manual pediatric fluid resuscitation (The "Push-Pull Technique" vs. the "Disconnect-Reconnect Technique") allows for the most rapid administration of normal saline when this is urgently required.

ELIGIBILITY:
Inclusion Criteria:

* Health Care Providers working or training at McMaster Children's Hospital, including staff nurses, staff physicians, postgraduate medical trainees, nursing students, and medical students
* may be asked to perform manual fluid resuscitation as part of their clinical care activities

Exclusion Criteria:

* Inability to understand English
* Limited manual dexterity, specifically resulting in an inability to perform manual fluid resuscitation involving syringes
* Have acted in a physically strenuous capacity that may result in significant hand fatigue in the 30 minutes immediately prior to performance of the intervention. Where this is the only criteria limiting subject participation, rescheduling of an alternate testing time will be permitted.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Overall fluid infusion rate | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Start Intervention Time is defined as the time that the model begins to effectively receive normal saline as administered by the participant, determined by the time at which fluid begins to collect in the graduated cylinder. End Intervention Time is defined as the time at which the model ceases to effectively receive further normal saline as determined by the time at which fluid stops collecting in the graduated cylinder. All testing will be videorecorded, with video reviews conducted by two independent and blinded outcome assessors using strict criteria to determine total intervention time (Total intervention time = end intervention time - start intervention time). At the time of subject testing, the research assistant will also record the total amount of normal saline collected in the graduated cylinder at the end of the intervention. Total intervention rate (mL/s) = volume of normal saline collected/Total intervention time.

SECONDARY OUTCOMES:
Accuracy of fluid volume delivery | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Total volume of normal saline (mL) effectively administered to the model by the participant
Catheter dislodgement event while performing the intervention | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Any IV catheter dislodgement events will be recorded by the research assistant at the time of subject testing on the data collection form. The IV catheter is transfixed to the hand of the mannequin in typical clinical fashion. The distal end of the catheter is located within conduit tubing which leads to a 1 litre graduated cylinder. Connected to the proximal aspect (hub) of the IV catheter is a 7 inch long IV Catheter Extension set, which the participant will be in contact with as they administer the intervention.
Self-reported fatigue | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Determined based upon responses to the study questionnaire which subjects will be asked to complete following performance of the intervention.
Fluid infusion rates for each of the three sequential fluid boluses | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Bolus 1 rate = 300 mL/Time to effectively administer the first 300 mL of fluid; Bolus 2 rate = 300 mL/Time to effectively administer the second 300 mL of fluid; Bolus 3 rate = Remaining volume effectively administered beyond the first 600 mL/Time to administer this remaining volume. Fluid administration times for Boluses 1, 2 and 3, will be determined based on video review in a similar fashion as for the Primary Outcome [Volume/(Bolus end time-Bolus start time)].

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Parker, MD, MSc, Principal Investigator — McMaster Children's Hospital
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Cole ET, Harvey G, Urbanski S, Foster G, Thabane L, Parker MJ. Rapid paediatric fluid resuscitation: a randomised controlled trial comparing the efficiency of two provider-endorsed manual paediatric fluid resuscitation techniques in a simulated setting. BMJ Open. 2014 Jul 3;4(7):e005028. doi: 10.1136/bmjopen-2014-005028. PMID 24993757
- [Derived] Cole ET, Harvey G, Foster G, Thabane L, Parker MJ. Study protocol for a randomised controlled trial comparing the efficiency of two provider-endorsed manual paediatric fluid resuscitation techniques. BMJ Open. 2013 Mar 21;3(3):e002754. doi: 10.1136/bmjopen-2013-002754. PMID 23524045
- See also: Protocol Publication — http://bmjopen.bmj.com/content/3/3/e002754.full.pdf